CLINICAL TRIAL: NCT06174545
Title: Effectiveness and Safety of Pigment Solution Program (PSP) as Adjuvant Therapy in Melasma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Collaborators: Menarini Group (Industry)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, SpKK(K), Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PSP
Record Dates: First submitted 2023-11-07; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (HQ group) (No Intervention): Group 1 is control group, getting SPF 30 sunscreen cream in the morning and only 2% Hydroquinone cream at night without a combination cream and facial soap that can be used in the morning and evening.
- Group 2 (PSP Group) (Experimental): Group 2, the treatment group, used PSP cleanser, PSP Day Cream and SPF 30 sunscreen in the morning and used Hydroquinone 2% and PSP Night Cream at night and PSP cleanser which was used in the morning and evening before using the cream.
  Interventions: Drug: Pigment Solution Program

INTERVENTIONS:
Drug: Pigment Solution Program — adjuvant therapy for melasma that contains of combination formula consisting of morning cream - containing kojic acid, Vitamin E, Vitamin A and AquaxylTM complex; night cream - contains kojic acid, glycolic acid and AquaxylTM complex, scrub granules; and cleaning fluid containing vegetable oil and lactic acid.
  Arms: Group 2 (PSP Group)

SUMMARY:
This research is a clinical study with a single-blind randomized clinical trial design (randomized controlled trial) in multicenters at two Dermatology and Venereology Education centers in Indonesia.

This study aims to determine the effectiveness and safety of PSP as adjuvant therapy for melasma.

This research will be attended by 33 research subjects

DETAILED DESCRIPTION:
Melasma is one of the most common hyperpigmentary dermatoses, found mostly in Asian or Hispanic people living in tropical areas.

The goal of melasma treatment is to remove existing pigmentation and to inhibit pigmentation. Until now, hydroquinone (HQ) is still used as the Gold Standard for melasma therapy.

Various epidemiological studies calculate the prevalence of melasma, it is estimated that the prevalence of melasma is 1% in the general population and in high risk populations it is 9 - 50%. This large variation is due to differences in skin type, ethnicity, and level of UV exposure

The diagnosis of melasma is based on the clinical picture, namely light to dark brown macules with irregular edges and a distribution that tends to be symmetrical, especially on the face. Supporting examinations can be carried out to determine the degree of melasma and monitor the therapy given.

This research is a clinical study with a single-blind randomized clinical trial design (randomized controlled trial) in multicenters at two Dermatology and Venereology Education centers in Indonesia. The number of samples was 33 divided into 2 groups based on consecutive sampling to obtain subjects who met the eligibility criteria. Then subjects will be allocated into two groups using block randomization.

What is meant by group 1 is control, getting SPF 30 sunscreen cream in the morning and only 2% Hydroquinone cream at night without a combination cream and facial soap that can be used in the morning and evening. Meanwhile, group 2, the treatment group, used PSP cleanser, PSP Day Cream and SPF 30 sunscreen in the morning and used Hydroquinone 2% and PSP Night Cream at night and PSP cleanser which was used in the morning and evening before using the cream.

Data collection and research will be carried out for 3 months and data management and analysis will be carried out for the following 1 month. Follow up will be carried out at Week 4, Week 8 and Week 12. Each follow up will be analyzed as follows:

* Physical examination
* 5 position face photos
* Mexameter examination
* Dermoscopic examination
* Check wood lamp
* MelasQoL check
* Calculation of mMASI Score
* Completing the Investigator's Global Assessment questionnaire
* Completing the Patient's Global Assessment Questionnaire
* Completing the Investigator's Tolerability Assessment questionnaire

Data is recorded in research status which is then compiled into a master table. After recording the research results is complete, the masking code is opened for statistical analysis. Data analysis used statistical tests in accordance with the intention to treat approach with research subject analysis methods based on intervention groups. The research results are attached in the form of narratives, frequency tables and graphs. The data will be processed statistically by a statistical consultant. Thus, data from SPs who dropped out will be included in the data analysis. The hypothesis test to assess changes in the primary end point (degree of melasma) during the study measurement series (baseline, M4, M8, M12) will be assessed using the Independent Sample T-test. Normality was tested using the Kolmogorov Smirnov normality test which was confirmed with the Coefficient of Variation. The data was processed statistically by a statistical consultant using SPSS® version 21.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 30-60 years
2. Fitzpatrick skin phototype IV-V
3. Diagnosis of epidermal, mixed and dermal types of Melasma

Exclusion Criteria:

1. Are pregnant or breastfeeding
2. Use other lightening agents, both oral and topical
3. Allergy to PSP content
4. Use of other topical therapies for skin disorders may interfere with the evaluation of melasma conditions
5. Suffering from other skin diseases such as acne, dermatitis
6. Using hormonal birth control

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 33 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-12-18 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Melasma Severity based on modified Melasma Severity Index (mMASI) score. | re-evaluation on day 28, day 56 and day 84 of therapy
  The range of values for mMASI is between 0 and 24 which can then be divided into mild melasma (0-8), moderate (8-16), and severe (16-24).
  The range of values for mMASI is between 0 and 24 which can then be divided into mild melasma (0-8), moderate (8-16), and severe (16-24).
  improvement occurs if the mMASI score decreases by <50% from the previous visit worsening if score persists or mMASI Score Increase >50%
Change of Melasma Severity based on Investigator Global Assesment (IGA). | re-evaluation on day 28, day 56 and day 84 of therapy
  Assessment of response to therapy as follows:
  * No effect: 0 (no visible change in Pigmentation)
  * Mild: 1 (decreased visible pigmentation, but still visible boundaries)
  * Moderate: 2 (obvious decrease in Pigmentation, but still limited visible)
  * Very good: 3 (disappearance of all visible abnormalities Pigmentation)
  improvement if there is >50% improvement from the previous visit worsening if score persists or improvement <50%
Change of Melasma Severity based on Investigator Tolerability Assesment (ITA). | re-evaluation on day 84 of therapy
  is one method of evaluating patient tolerability of products which is assessed subjectively by investigators.
  Assessment of patient tolerability as follows:
  * 0 = no tolerability,
  * 1 = moderate tolerability,
  * 2 = good tolerability,
  * 3 = very good tolerability.
  tolerability was good if the score improved >50% from the previous visit worsening if score persists or improvement <50%
Change of Melasma Severity based on Patient's Tolerability Assesment (PtGA). | re-evaluation on day 28, day 56 and day 84 of therapy
  one method of evaluating the response to therapy in melasma which is assessed subjectively by the patient. The response to therapy can be assessed as follows
  * No or slight response: < 25% improvement
  * Moderate response: 25% - 50% improvement
  * Good response: 50% improvement - < 75%
  * Excellent response: improvement > 75%
  The response is said to be good if the score is above 50% since the previous visit
Change of Melanin and Erythema Index Based on Mexameter | re-evaluation on day 28, day 56 and day 84 of therapy
  improves if there is a decrease in melanin levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in melanin levels or there is a decrease of <50%
Change of Melasma Severity based on Dermoscopy | re-evaluation on day 84 of therapy
  based on Dermoscopy
  Telangiectasis score assessment using a 5-point dermoscopy-scale:
  0 = No visible capillaries.
  1 = Elongated capillaries accompanied by dilation, not visible to the naked eye. 2 = Moderate telangiectasis that is beginning to be visible to the naked eye.
  3 = Severe telangiectasis characterized by reduced capillary loops. 4 = Very severe telangiectasis characterized by dilatation and loss of capillary loops.
Change of Melasma Severity based on Wood's Lamp | re-evaluation on day 84 of therapy
  Epidermal Type/ Dermal Typed/ Mixed Typed
Compare Quality Of Life based on MelasQoL Score | re-evaluation on day 84 of therapy
  based on MelasQoL Score minimum score: 7 maximum score : 70

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Umum Pusat Nasional Dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided